CLINICAL TRIAL: NCT05238103
Title: Impact of a Mobile Technology Enabled Corrie Cardiac Rehabilitation Program on Functional Status and Cardiovascular Outcomes (mTECH-Rehab): A Randomized Controlled Trial
Brief Title: Impact of a Corrie Cardiac Rehabilitation Program
Acronym: mTECH-Rehab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: American Heart Association (Other); Apple Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00308410
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Results first posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Disease; Myocardial Infarction; Myocardial Ischemia; Coronary Artery Occlusion; Coronary Artery Stenosis Stent; Bypass Graft Occlusion; Valve Heart Disease
Keywords: digital health; smartphone app; self-management; guideline adherence; behavior modification; community engagement
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction; Myocardial Ischemia; Coronary Occlusion; Heart Valve Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) (Experimental): Receives Corrie Virtual Cardiac Rehabilitation Program along with option to continue traditional, center-based cardiac rehabilitation.
  Interventions: Combination Product: Corrie Hybrid Cardiac Rehabilitation Program
- Facilitated Center-Based Cardiac Rehabilitation Program (Control Group) (No Intervention): Receives traditional, center-based cardiac rehabilitation. The study team will help facilitate the logistics of receiving center-based cardiac rehabilitation, including proper referrals.

INTERVENTIONS:
Combination Product: Corrie Hybrid Cardiac Rehabilitation Program — The Corrie Hybrid Cardiac Rehabilitation Program is a multi-component intervention. It consists of the Corrie smartphone app for cardiovascular health optimization which is paired with wristband device (Apple Watch or Fitbit), Bluetooth-enabled Omron blood pressure monitor and exercise resistance bands. The program also includes individualized treatment plan development, setting health goals and communication with trained Corrie Health Coach. Furthermore, the intervention includes motivational text messages sent to participants throughout the study to aid with risk factor modification.
  Arms: Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group)

SUMMARY:
In this randomized clinical trial, the researchers are investigating whether a multi-component virtual/hybrid cardiac rehabilitation program will improve functional status, cholesterol level, overall cardiovascular health, individual risk factors, quality of life and mental health for patients who have recently been diagnosed with myocardial infarction, received a coronary stent, underwent heart surgery or catheter-based valve replacement, as compared to traditional, center-based cardiac rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Individuals admitted to the hospital for the following conditions or interventions during the index admission: Acute myocardial infarction (STEMI or NSTEMI type 1), Coronary artery bypass grafting (CABG), and Coronary artery angioplasty/stenting (PCI), Heart valve surgery, catheter-based aortic valve replacement (TAVR).

Exclusion Criteria

* Non-English speaking
* Symptomatic severe aortic stenosis or other severe valvular disease
* Physical disability that would preclude safe and adequate exercise performance
* Hypertrophic obstructive cardiomyopathy with peak resting left ventricular outflow gradient of >25 mmHg
* Known aortic dissection
* Severe resting arterial hypertension (Systolic blood pressure >200 mmHg or diastolic BP >110mmHg) at baseline assessment
* Mental impairment leading to inability to cooperate with study procedures
* Untreated high degree atrioventricular block
* Atrial fibrillation with uncontrolled ventricular rate (Heart rate >110 at rest) at baseline assessment
* History of cardiac arrest or sudden death
* Myocardial infarction or cardiac surgery complications with cardiogenic shock and/or congestive heart failure and/or signs/symptoms of post-procedure ischemia
* Left ventricular ejection fraction <40%
* History of Clinically significant depression
* Visual or hearing impairment which precludes the use of the intervention
* Presence of cardiac defibrillator
* Incomplete revascularization procedure
* History of one or more episodes of falls in the last year
* Pregnancy

  * If patients are deemed clinically unstable and unable to participate at the time of initial screening, the research team member may return at a later date to determine whether this status has changed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2024-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lena Mathews, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified, aggregate level results, including primary and secondary outcomes, and the data dictionary will be shared through clinicaltrials.gov. Study documents (study protocol, statistical analysis plan, informed consent form, analytic code) will also be shared upon request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: IPD will be made available upon request for up to 3 years from the study completion date (to 10/14/2027).
Access Criteria: Researchers must submit a letter of intention and formal data request to the mTECH-Rehab principal investigator, who will review the request with the core study team and grant approval based on evaluation of merit.
URL: https://clinicaltrials.gov/policy/protocol-definitions?popup=true#ipd-sharing

REFERENCES:
- [Background] Isakadze N, Kim CH, Marvel FA, Ding J, MacFarlane Z, Gao Y, Spaulding EM, Stewart KJ, Nimbalkar M, Bush A, Broderick A, Gallagher J, Molello N, Commodore-Mensah Y, Michos ED, Dunn P, Hanley DF, McBee N, Martin SS, Mathews L. Rationale and Design of the mTECH-Rehab Randomized Controlled Trial: Impact of a Mobile Technology Enabled Corrie Cardiac Rehabilitation Program on Functional Status and Cardiovascular Health. J Am Heart Assoc. 2024 Jan 16;13(2):e030654. doi: 10.1161/JAHA.123.030654. Epub 2024 Jan 16. PMID 38226511

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Assessed for eligibility: 6,170; Met eligibility criteria: 1,252; Met exclusion criteria: 4,918; Excluded: 993 (Declined to participate: 710, Unable to be contacted: 283).
Pre-assignment Details: Drop-out (pre-randomization/run-in) - 57. (Lost to follow up - 32. Developed exclusion criteria -10. Withdrew consent - 8. Financial reason - 5. Unable to undergo safety evaluation - 2). 259 Enrolled. 202 participants randomized.
Period: Overall Study
Arm/Group | Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) | Facilitated Center-Based Cardiac Rehabilitation Program (Control Group)
Started | 101 | 101
Completed | 85 | 77
Not Completed | 16 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) | Facilitated Center-Based Cardiac Rehabilitation Program (Control Group) | Total
Number analyzed (Participants) | 101 | 101 | 202
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.6 (12.4) | 63.3 (11.5) | 63.9 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 32 | 65
  Male | 68 | 69 | 137
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 83 | 82 | 165
  African American | 8 | 10 | 18
  Asian | 6 | 5 | 11
  Hispanic or Latino | 0 | 2 | 2
  Other | 3 | 2 | 5
  Declined to answer | 1 | 0 | 1
Cardiac Rehabilitation Indication (Disease Category + Treatment Modality) [Count of Participants; unit: Participants] — AMI: Acute myocardial infarction, CAD: Coronary artery disease, CABG: Coronary artery bypass grafting surgery, PCI: Percutaneous coronary intervention, TAVR: Transcatheter aortic valve replacement, VHD: Valvular heart disease
  Participants
    AMI (Medically treated) | 0 | 1 | 1
    AMI (Treated with PCI) | 15 | 18 | 33
    AMI (Treated with CABG) | 2 | 1 | 3
    CAD without AMI (Treated with PCI) | 29 | 30 | 59
    CAD without AMI (Treated with CABG) | 15 | 11 | 26
    VHD (Treated with TAVR) | 10 | 3 | 13
    VHD (Treated with Heart valve surgery) | 27 | 35 | 62
    Combined CABG + Heart valve surgery | 3 | 2 | 5
Clinical History [Count of Participants; unit: Participants] — Participants may fit into more than one category
  Participants
    Hypertension | 76 | 77 | 153
    Hyperlipidemia | 83 | 88 | 171
    Diabetes mellitus | 25 | 19 | 44
    Tobacco use | 2 | 2 | 4
    Coronary artery disease | 75 | 80 | 155
    Myocardial infarction | 30 | 32 | 62
    Atrial fibrillation | 38 | 28 | 66
    Valvular heart disease | 43 | 42 | 85
    Heart failure | 15 | 18 | 33
Cardiac Rehabilitation Indication (Disease Category) [Count of Participants; unit: Participants] — AMI: Acute myocardial infarction, CAD: Coronary artery disease, CABG: Coronary artery bypass grafting surgery, PCI: Percutaneous coronary intervention, TAVR: Transcatheter aortic valve replacement, VHD: Valvular heart disease
  Participants
    AMI | 17 | 20 | 37
    CAD without AMI | 44 | 41 | 85
    VHD | 37 | 38 | 75
    CAD with VHD | 3 | 2 | 5
Blood Pressure (mmHg) [Mean (Standard Deviation); unit: mmHg]
  Systolic blood pressure (mmHg) | 124.3 (16.1) | 126.8 (17.3) | 125.3 (16.7)
  Diastolic blood pressure (mmHg) | 70.7 (9.8) | 70.9 (10.5) | 70.8 (10.1)
Heart Rate (beats per minute) [Mean (Standard Deviation); unit: beats per minute] | 74.2 (12.7) | 73.1 (12.6) | 73.6 (12.6)
Weight (kilograms) [Mean (Standard Deviation); unit: kilograms] | 90.8 (21.5) | 84.6 (16.2) | 87.7 (19.3)
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 29.7 (6.0) | 28.5 (5.3) | 29.1 (5.7)
Left Ventricular ejection fraction (LVEF) [Mean (Standard Deviation); unit: Percentage of LVEF] | 58.2 (7.7) | 59.2 (6.7) | 58.7 (7.2)

OUTCOME MEASURES:

1. Secondary Outcome: Composite Cardiovascular Health Metric for Secondary Prevention
Description: The cardiovascular health metric for secondary prevention (adapted from American Heart Association's Life Simple 7). The score ranges from 0 to 14 with higher score indicating better cardiovascular health.
Time Frame: 12 weeks after randomization
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) | Facilitated Center-Based Cardiac Rehabilitation Program (Control Group)
Number analyzed (Participants) | 101 | 101
Score on a scale | 9.6 (1.7) | 9.5 (1.7)
Statistical Analysis 1: Comparison: Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) vs Facilitated Center-Based Cardiac Rehabilitation Program (Control Group); Test type: Superiority; p = 0.58, t-test, 2 sided

2. Secondary Outcome: Blood Pressure (mmHg)
Description: Systolic blood pressure and Diastolic blood pressure
Time Frame: 12 weeks after randomization
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) | Facilitated Center-Based Cardiac Rehabilitation Program (Control Group)
Number analyzed (Participants) | 101 | 101
mmHg
  Systolic blood pressure | 122.7 (13.8) | 121.0 (13.6)
  Diastolic blood pressure | 70.5 (11.5) | 68.6 (10.8)
Statistical Analysis 1: Comparison: Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) vs Facilitated Center-Based Cardiac Rehabilitation Program (Control Group); For systolic blood pressure; Test type: Superiority; p = 0.40, t-test, 2 sided
Statistical Analysis 2: Comparison: Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) vs Facilitated Center-Based Cardiac Rehabilitation Program (Control Group); For diastolic blood pressure; Test type: Superiority; p = 0.25, t-test, 2 sided

3. Secondary Outcome: Low Density Lipoprotein - Cholesterol (LDL-C)
Description: LDL cholesterol level (in mg/dl) measured through blood sample drawn at 12 week follow up visit
Time Frame: 12 weeks after randomization
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) | Facilitated Center-Based Cardiac Rehabilitation Program (Control Group)
Number analyzed (Participants) | 101 | 101
mg/dL | 65.6 (33.1) | 71.4 (31.4)
Statistical Analysis 1: Comparison: Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) vs Facilitated Center-Based Cardiac Rehabilitation Program (Control Group); Test type: Superiority; p = 0.27, t-test, 2 sided

4. Secondary Outcome: Glycosylated Hemoglobin (HbA1c)
Description: Glycosylated hemoglobin (HbA1c) level (%) measured through blood sample drawn at 12 week follow up visit
Time Frame: 12 weeks after randomization
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) | Facilitated Center-Based Cardiac Rehabilitation Program (Control Group)
Number analyzed (Participants) | 101 | 101
percentage of glycated hemoglobin | 5.8 (0.7) | 5.9 (0.8)
Statistical Analysis 1: Comparison: Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) vs Facilitated Center-Based Cardiac Rehabilitation Program (Control Group); Test type: Superiority; p = 0.39, t-test, 2 sided

5. Secondary Outcome: Body Mass Index (kg/m^2)
Description: BMI = weight (kg) / height in meters squared (m^2). Weight and height measured by study staff at study visit.
Time Frame: 12 weeks after randomization
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) | Facilitated Center-Based Cardiac Rehabilitation Program (Control Group)
Number analyzed (Participants) | 101 | 101
kg/m^2 | 30.2 (6.7) | 28.7 (7.4)
Statistical Analysis 1: Comparison: Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) vs Facilitated Center-Based Cardiac Rehabilitation Program (Control Group); Test type: Superiority; p = 0.19, t-test, 2 sided

6. Secondary Outcome: Quality of Life as Assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health-10
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health-10: The 10-item patient-reported questionnaire administered at 12 weeks follow up in which the response options are presented as 5-point (as well as a single 11-point) rating scales. The results of the questions are used to calculate two summary scores: a Global Physical Health Score and a Global Mental Health score. These scores are then standardized to the general population, using the "T-Score". The average "T-Score" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient.
Time Frame: 12 weeks after randomization
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) | Facilitated Center-Based Cardiac Rehabilitation Program (Control Group)
Number analyzed (Participants) | 101 | 101
t-score
  Global physical health score | 50.4 (7.4) | 52.0 (6.9)
  Global mental health score | 52.0 (8.4) | 52.1 (7.4)
Statistical Analysis 1: Comparison: Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) vs Facilitated Center-Based Cardiac Rehabilitation Program (Control Group); For: Global physical health score; Test type: Superiority; p = 0.16, t-test, 2 sided
Statistical Analysis 2: Comparison: Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group); For: Global mental health score; Test type: Superiority; p = 0.71, t-test, 2 sided

7. Secondary Outcome: Blood Pressure Control
Description: Blood pressure control (Cardiovascular secondary health metric component). Ideal (SBP <130 mmHg and DBP <90 mmHg). Intermediate (SBP 130-139 mmHg or DBP 80-89 mmHg). Poor (SBP ≥140 mmHg or DBP ≥90 mmHg).
Time Frame: 12 weeks after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) | Facilitated Center-Based Cardiac Rehabilitation Program (Control Group)
Number analyzed (Participants) | 101 | 101
Participants
  Ideal | 59 | 65
  Intermediate | 34 | 27
  Poor | 8 | 9
Statistical Analysis 1: Comparison: Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) vs Facilitated Center-Based Cardiac Rehabilitation Program (Control Group); Test type: Superiority; p = 0.60, Chi-squared

8. Secondary Outcome: Cholesterol (LDL-C) Control
Description: Cholesterol (LDL-C) control (Cardiovascular secondary health metric component). Ideal (LDL-C <70mg/dL). Intermediate (LDL-C 70-99 mg/dL). Poor (LDL-C ≥100mg/dL)
Time Frame: 12 weeks after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) | Facilitated Center-Based Cardiac Rehabilitation Program (Control Group)
Number analyzed (Participants) | 101 | 101
Participants
  Ideal | 62 | 52
  Intermediate | 23 | 30
  Poor | 16 | 19
Statistical Analysis 1: Comparison: Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) vs Facilitated Center-Based Cardiac Rehabilitation Program (Control Group); Test type: Superiority; p = 0.57, Chi-squared

9. Secondary Outcome: Diabetes Control
Description: Diabetes (HbA1c) control (Cardiovascular secondary health metric component). Ideal (HbA1c <7% for diabetic, <5.7% for non-diabetic). Intermediate (HbA1c 7.0-7.9% for diabetic, 5.0-5.9% for non-diabetic). Poor (HbA1c ≥8% for diabetic, ≥6.5% for non-diabetic).
Time Frame: 12 weeks after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) | Facilitated Center-Based Cardiac Rehabilitation Program (Control Group)
Number analyzed (Participants) | 101 | 101
Participants
  Ideal | 66 | 55
  Intermediate | 32 | 40
  Poor | 3 | 6
Statistical Analysis 1: Comparison: Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) vs Facilitated Center-Based Cardiac Rehabilitation Program (Control Group); Test type: Superiority; p = 0.28, Chi-squared

10. Secondary Outcome: Weight (BMI) Categories
Description: Weight (BMI) categories (Cardiovascular secondary health metric component). Ideal (BMI <25 kg/m^2). Intermediate (BMI 25-29 kg/m^2). Poor (BMI ≥ 30 kg/m^2).
Time Frame: 12 weeks after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) | Facilitated Center-Based Cardiac Rehabilitation Program (Control Group)
Number analyzed (Participants) | 101 | 101
Participants
  Ideal | 25 | 29
  Intermediate | 23 | 35
  Poor | 53 | 37
Statistical Analysis 1: Comparison: Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) vs Facilitated Center-Based Cardiac Rehabilitation Program (Control Group); Test type: Superiority; p = 0.09, Chi-squared

11. Secondary Outcome: Physical Activity Categories
Description: Physical activity categories (Cardiovascular secondary health metric component). Ideal (≥150 min/wk moderate physical activity, ≥75 min/wk vigorous physical activity). Intermediate (1-149 min/wk moderate physical activity, 1-74 min/wk vigorous physical activity). Poor (No regular exercise).
Time Frame: 12 weeks after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) | Facilitated Center-Based Cardiac Rehabilitation Program (Control Group)
Number analyzed (Participants) | 101 | 101
Participants
  Ideal | 72 | 81
  Intermediate | 29 | 18
  Poor | 0 | 2
Statistical Analysis 1: Comparison: Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) vs Facilitated Center-Based Cardiac Rehabilitation Program (Control Group); Test type: Superiority; p = 0.19, Chi-squared

12. Secondary Outcome: Diet Categories
Description: Diet categories (Cardiovascular secondary health metric component). Ideal (Rate Your Plate score 64-81). Intermediate (Rate Your Plate score 46-63). Poor (Rate Your Plate score 27-45).
Time Frame: 12 weeks after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) | Facilitated Center-Based Cardiac Rehabilitation Program (Control Group)
Number analyzed (Participants) | 101 | 101
Participants
  Ideal | 62 | 57
  Intermediate | 39 | 44
  Poor | 0 | 0
Statistical Analysis 1: Comparison: Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) vs Facilitated Center-Based Cardiac Rehabilitation Program (Control Group); Test type: Superiority; p = 0.60, Chi-squared

13. Secondary Outcome: Tobacco Use
Description: Tobacco use categories (Cardiovascular secondary health metric component). Ideal (never). Intermediate (Former smoker). Poor (Recent/Current smoker).
Time Frame: 12 weeks after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) | Facilitated Center-Based Cardiac Rehabilitation Program (Control Group)
Number analyzed (Participants) | 101 | 101
Participants
  Ideal/Intermediate (Never/Former smoker) | 99 | 89
  Poor (Recent/Current smoker) | 2 | 12
Statistical Analysis 1: Comparison: Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) vs Facilitated Center-Based Cardiac Rehabilitation Program (Control Group); Test type: Superiority; p = 1.00, Chi-squared

14. Secondary Outcome: Cardiac Rehabilitation Engagement
Description: Cardiac rehabilitation engagement as measured by number of participants who attended the sessions per category. Grouped by Healthcare Effectiveness Data and Information Set (HEDIS) categories: Initiation (0-12 sessions attended), Engagement 1 (13-24 sessions attended), Engagement 2 (25-36 sessions attended).
Time Frame: 12 weeks after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) | Facilitated Center-Based Cardiac Rehabilitation Program (Control Group)
Number analyzed (Participants) | 101 | 101
Participants
  Initiation (0-12 sessions attended) | 37 | 31
  Engagement 1 (13-24 sessions attended) | 20 | 29
  Engagement 2 (25-36 sessions attended) | 44 | 41
Statistical Analysis 1: Comparison: Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) vs Facilitated Center-Based Cardiac Rehabilitation Program (Control Group); Test type: Superiority; p = 0.35, Chi-squared

15. Other Pre Specified Outcome: Depression as Assessed by the Patient Health Questionnaire 8
Description: The difference in depressive symptoms as measured by Patient Health Questionnaire 8 (PHQ 8): The 8 item questionnaire administered at 12 weeks with the following scoring system: Score range 0-24. A score of 10 or greater is considered major depression, 20 or more is severe major depression.
  Note, as an exploratory outcome, only a subgroup of participants responded to this survey request.
Time Frame: 12 weeks after randomization
Population: Note, as an exploratory outcome, only a subgroup of randomized study participants responded to this survey request.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) | Facilitated Center-Based Cardiac Rehabilitation Program (Control Group)
Number analyzed (Participants) | 79 | 66
score on a scale | 2 [0 to 5] | 2 [0 to 4]

16. Other Pre Specified Outcome: Anxiety as Assessed by the Generalized Anxiety Disorder 7
Description: The difference in anxiety level as measured by Generalized Anxiety Disorder 7 (GAD 7): The 7-item questionnaire administered at 12 weeks follow up with the following scoring system. Each item is assigned scores of 0, 1, 2, and 3 to the response categories. GAD-7 total score for the seven items ranges from 0 to 21. 0-4: minimal anxiety 5-9: mild anxiety 10-14: moderate anxiety 15-21: severe anxiety.
Time Frame: 12 weeks after randomization
Population: Note, as an exploratory outcome, only a subgroup of randomized study participants responded to this survey request.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) | Facilitated Center-Based Cardiac Rehabilitation Program (Control Group)
Number analyzed (Participants) | 79 | 66
score on a scale | 1 [0 to 4] | 1 [0 to 4]

17. Other Pre Specified Outcome: Stress as Assessed by the Perceived Stress Scale-10
Description: The difference in stress level as measured by Perceived Stress Scale (PSS -10): The 10 item questionnaire administered at 12 weeks follow up. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
Time Frame: 12 weeks after randomization
Population: Note, as an exploratory outcome, only a subgroup of randomized study participants responded to this survey request.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) | Facilitated Center-Based Cardiac Rehabilitation Program (Control Group)
Number analyzed (Participants) | 79 | 66
Score on a scale | 11.5 (6.6) | 11.0 (6.9)

18. Other Pre Specified Outcome: Health Literacy as Assessed by the (e) Health Literacy Scale (eHEALS)
Description: The difference in Health Literacy as measured by The (e) Health Literacy Scale (eHEALS): The 8 item scale administered at 12 weeks follow up. Total scores of the eHEALS range from 8 to 40, with higher scores representing higher self-perceived (e) Health literacy.
Time Frame: 12 weeks after randomization
Population: Note, as an exploratory outcome, only a subgroup of randomized study participants responded to this survey request.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) | Facilitated Center-Based Cardiac Rehabilitation Program (Control Group)
Number analyzed (Participants) | 80 | 69
Score on a scale | 31.7 (5.5) | 32.3 (5.1)

19. Other Pre Specified Outcome: Patient Activation as Assessed by the Patient Activation Measure 10
Description: The difference in patient activation as measured by Patient Activation Measure 10 (PAM 10): The 10-item five-point Likert scale for assessing patient activation at 12 weeks follow up, indicating whether the patient possesses the necessary knowledge, skills, and confidence needed for self-care. The total score reference range is from 0 to 100, where higher scores indicate greater patient activation and ability for self-care.
Time Frame: 12 weeks after randomization
Population: Note, as an exploratory outcome, only a subgroup of randomized study participants responded to this survey request.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) | Facilitated Center-Based Cardiac Rehabilitation Program (Control Group)
Number analyzed (Participants) | 80 | 69
Score on a scale | 33.7 (4.7) | 35.1 (3.4)

20. Primary Outcome: 6-minute Walking Distance (Meters)
Description: Mean difference in 6 minute walk distance, between Intervention and Control groups, as measured at final study visit occurring at 12 weeks after randomization.
Time Frame: 12 weeks after randomization
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) | Facilitated Center-Based Cardiac Rehabilitation Program (Control Group)
Number analyzed (Participants) | 101 | 101
meters | 506.1 (113.9) | 489.8 (104.0)
Statistical Analysis 1: Comparison: Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) vs Facilitated Center-Based Cardiac Rehabilitation Program (Control Group); Significance testing: Generalized regression model; Test type: Non-Inferiority — The non-inferiority margin of 12.5 meters was chosen to represent about 40% of the minimum important difference of 30 meters in the 6 minute walk test as identified in previous studies. For sample size calculation, to allow for an attrition rate of 20% during follow up after randomization, a total of 200 (100 per group) participants were needed to be recruited and then randomized in a 1:1 ration to Intervention vs. Control groups; p = 0.04, t-test, 1 sided; Mean Difference (Final Values) = 16.3, 95% CI 1-sided [lower limit -9.1]

21. Other Pre Specified Outcome: User Engagement as Assessed by the Number of App Interactions (Intervention Group Only)
Description: Number of interactions in the smartphone app per participant, collected via the Corrie Health Platform User Analytics at 12 weeks follow up (only assessed in intervention arm).
Time Frame: 12 weeks after randomization
Measure: Mean (Standard Deviation); unit: app interactions
Arm/Group | Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group)
Number analyzed (Participants) | 101
app interactions
  App interaction for heart rate event | 11821.6 (17364.7)
  App interaction for blood pressure event | 16.9 (19.0)
  App interaction for exercise completion event | 34.9 (38.7)
  App interaction for medication taken event | 296.5 (264.7)
  App interaction for weight check event | 51.7 (35.9)
  App interaction for mood check event | 53.7 (35.6)
  App interaction for step count check event | 125.7 (168.9)
  App interaction for education event | 17.7 (8.4)

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up at 12 weeks after randomization
Description: Reported mortality (by electronic health record review or family report), serious adverse events (by electronic health record review or family report), or minor events (by patient report)
Arm/Group | Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) | Facilitated Center-Based Cardiac Rehabilitation Program (Control Group)
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/101
Serious Adverse Events (participants affected / at risk) | 2/101 | 9/101
Other Adverse Events (participants affected / at risk) | 4/101 | 2/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) (N=101) | Facilitated Center-Based Cardiac Rehabilitation Program (Control Group) (N=101)
Acute decompensated heart failure (Cardiac disorders) | 1 (1) | 0 (0) — Acute decompensated heart failure requiring hospitalization
Atrial fibrillation with rapid ventricular response (Cardiac disorders) | 1 (1) | 0 (0) — Atrial fibrillation with rapid ventricular response requiring hospitalization
ST-elevation myocardial infarction (STEMI) due to bypass graft occlusion (Cardiac disorders) | 0 | 1 — ST-elevation myocardial infarction (STEMI) due to bypass graft occlusion requiring hospitalization
Stress cardiomyopathy (Cardiac disorders) | 0 | 1 — Stress cardiomyopathy requiring hospitalization
Syncope (Nervous system disorders) | 0 | 1 — Syncope event requiring hospitalization
Chest pain (non-cardiac) (Musculoskeletal and connective tissue disorders) | 0 | 2 — Non-cardiac chest pain requiring hospitalization
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 2 — Gastrointestinal disorder requiring hospitalization
Infection (Infections and infestations) | 0 | 2 — Infection requiring hospitalization
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Corrie Hybrid Cardiac Rehabilitation Program (Intervention Group) (N=101) | Facilitated Center-Based Cardiac Rehabilitation Program (Control Group) (N=101)
Symptoms during 6 minute walk test (Musculoskeletal and connective tissue disorders) | 2 | 1 — Patient reporting significant symptoms during 6 minute walk test requiring early termination or modification of 6MWT protocol
Chest pain at home (non-cardiac) (Musculoskeletal and connective tissue disorders) | 1 | 0 — Chest pain at home, deemed non-cardiac etiology and not requiring hospitalization
Pain from wearable device (Musculoskeletal and connective tissue disorders) | 1 | 0 — Significant pain from wearable device, precluding meaning use of technology and hybrid CR intervention
Delayed blood sample processing (Product Issues) | 0 | 1 — Delayed blood sample processing for lab sample collected during final study visit

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-09): https://cdn.clinicaltrials.gov/large-docs/03/NCT05238103/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-27): https://cdn.clinicaltrials.gov/large-docs/03/NCT05238103/ICF_001.pdf